CLINICAL TRIAL: NCT00996151
Title: A Healthy Volunteer, Single Dose Phase I Trial to Determine the Amount of Testerone MD-Lotion 2% Remaining on the Axilla After Washing.
Brief Title: Testosterone MD-Lotion Residual Washing Study
Acronym: MTE11
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrux DDS Pty Ltd (Industry)
Responsible Party: Tina Soulis, Director, Clinical Development, Acrux Pharma Pty Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MTE11
Record Dates: First submitted 2009-10-12; First posted 2009-10-16 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Hypergonadism
Keywords: Hypergonadism; Testosterone Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Testosterone MD-Lotion — Single dose Testosterone MD-Lotion 2%

SUMMARY:
The study will evaluate the amount of Testosteron MD-Lotion 2% remaining on the axilla after a single dose application in healthy males who undergo a post dose washing procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects ≥18 and ≤ 70 years

Exclusion Criteria:

* Disqualifying concurrent condition or allergy/sensitivity to Testosterone MD-Lotion

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The amount of Testerone MD-Lotion 2% remaining on the axilla after a single dose application in healthy males who undergo a post dose washing procedure. | March 2010

SECONDARY OUTCOMES:
The safety and tolerability of Testosterone MD-Lotion 2% following a single dose application. This will be performed by review of adverse events, EKG and assessment of laboratory parameters (haematology, biochemistry, urinalysis and hormone levels). | March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, PhD, Study Director — Acrux Pharma Pty Ltd
Locations (1):
- QPharm Pty Ltd, Brisbane, Queensland, Australia